CLINICAL TRIAL: NCT03693105
Title: A Multi-Site, Randomized, Double-Blind Trial Assessing The Effects of SAINT® Neuromodulation System on Explicit and Implicit Suicidal Cognition
Brief Title: The Effects of SAINT® Neuromodulation System on Explicit and Implicit Suicidal Cognition
Acronym: SAINT®SC
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Funding discontinued.
Sponsor: Magnus Medical (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLN-0105; R01MH125160 (NIH)
Record Dates: First submitted 2018-09-27; First posted 2018-10-02 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder; Major Depressive Episode; Suicidal Ideation
Keywords: Suicidality; Neuromodulation; Transcranial magnetic stimulation; Depression; Intermittent theta burst stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Suicidal Ideation; Depression

STUDY DESIGN:
Intervention Model Description: Patients will receive either active or sham stimulation to the DLPFC. Patients will be randomized to either condition with a 50:50 chance.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SAINT stimulation (Active Comparator): Active SAINT stimulation will be applied to the left dorsolateral prefrontal cortex (DLPFC)
  Interventions: Device: Active SAINT Stimulation
- Sham stimulation (Sham Comparator): Sham (non-active) stimulation will be applied to the left dorsolateral prefrontal cortex (DLPFC)
  Interventions: Device: Sham SAINT Stimulation

INTERVENTIONS:
Device: Active SAINT Stimulation — Participants who are randomly assigned to this group will receive active SAINT targeted to the left DLPFC. Stimulation intensity will be standardized at 90% of resting motor threshold (adjusted for cortical depth).
  Stimulation will be delivered using the Magventure Magpro X100 TMS system with the Cool-B65 A/P coil.
  Arms: SAINT stimulation
Device: Sham SAINT Stimulation — Participants who are randomly assigned to this group will receive sham stimulation targeted to the left DLPFC.
  Sham stimulation will be delivered using the Magventure Magpro X100 TMS system with the Cool-B65 A/P coil.
  Arms: Sham stimulation

SUMMARY:
This multi-site, double-blind, randomized, sham-controlled mechanistic trial aims to test the effects of Magnus Neuromodulation System (MNS) with Stanford Accelerated Intermittent Neuromodulation Therapy (SAINT®) Technology on the neural circuitry of suicidal cognitions in psychiatrically hospitalized patients with Major Depressive Disorder (MDD) and active suicidal ideation (SI). This will be accomplished by applying the MNS with SAINT to a customized target within the left dorsolateral prefrontal cortex (L-DLPFC) identified with fMRI for five consecutive days and measuring resting-state functional connectivity (RS FC) between the subgenual anterior cingulate cortex (sgACC) and the default mode network (DMN) at baseline and immediate-post visit. The relationship between changes in RS FC and changes in both Explicit and Implicit Suicidal Cognitions (ESC and ISC, respectively) will be determined. This study will also determine the relationship between changes in RS FC in neural networks underlying mediators of suicidal cognitions and changes in such mediators with active versus sham SAINT.

DETAILED DESCRIPTION:
This multi-site, double-blind, randomized, sham-controlled mechanistic trial aims to test the effects of Magnus Neuromodulation System (MNS) with Stanford Accelerated Intermittent Neuromodulation Therapy (SAINT®) Technology on the neural circuitry of suicidal cognitions in psychiatrically hospitalized patients with Major Depressive Disorder (MDD) and active suicidal ideation (SI). This will be accomplished by applying the MNS with SAINT protocol (10 applications per day to a customized target within the left dorsolateral prefrontal cortex (L-DLPFC) identified with fMRI for five consecutive days) and measuring resting-state functional connectivity (RS FC) between the subgenual anterior cingulate cortex (sgACC) and the default mode network (DMN) at baseline and immediate-post visit. The relationship between changes in RS FC and changes in both Explicit and Implicit Suicidal Cognitions (ESC and ISC, respectively) will be determined. This study will also determine the relationship between changes in RS FC in neural networks underlying mediators of suicidal cognitions and changes in such mediators (i.e., depression, hopelessness, anhedonia) with active versus sham SAINT.

The mechanistic hypothesis is that active SAINT modulates RS FC underlying ESC (sgACC-DMN) and ISC (DLPFC-ACC) and that these changes in connectivity will correlate with reductions in ESC and ISC, respectively. MDD with current Major Depressive Episode will be defined according to DSM-5 criteria, and active SI will be defined by a baseline modified Scale for Suicide Ideation (M-SSI) score ≥ 9.

The primary objective is to determine if active versus sham SAINT aiTBS applied to the left dorsolateral prefrontal cortex (L-DLPFC)-subgenual anterior cingulate cortex (sgACC) is effective in modulating neural networks underlying explicit suicidal cognition (ESC) in psychiatric inpatients.

The secondary objective is to determine if active versus sham SAINT aiTBS applied to the L-DLPFC-sgACC is effective in modulating neural networks underlying implicit suicidal cognition (ISC) in psychiatric inpatients.

The tertiary objective is to determine if active versus sham SAINT aiTBS applied to the L-DLPFC-sgACC is effective in modulating neural networks underlying mediators of suicidal cognitions such as depression, hopelessness, and anhedonia.

The study will enroll approximately 100 participants and employ a two-arm design with 50 subjects per arm. The target population is adults of all genders and ethnicities who are between 18 and 75 years of age with a diagnosis of treatment-resistant MDD experiencing a current Major Depressive Episode, with active suicidal ideation, and who are otherwise in good general health. Participants must be without contraindications to Magnetic Resonance Imaging (MRI) or transcranial magnetic stimulation (TMS) and must be able to attend all study visits.

This study will deliver both active and sham SAINT via a MagPro X100 edition (MagVenture, Skovlunde, Denmark) TMS device equipped with a Cool-B65 A/P coil. The stimulation paradigm consists of 10 daily sessions (50 total over 5-days) of MNS with SAINT stimulation (3-pulse 50-Hz bursts at 5-Hz for 2-second trains, with trains every 10 seconds), delivered with 50-minute inter-session intervals (10-minute sessions, 50-minutes in between sessions). Stimulation will be delivered at 90% of the resting motor threshold (with depth correction to account for the distance between the scalp and cortex). An operator entered code (derived from the study EDC) will instruct the device to deliver active or sham magnetic stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of all genders between the ages of 18 and 75 years at the time of screening.
2. Able to read, understand, and provide written, dated informed consent prior to screening.
3. Proficiency in English sufficient to complete questionnaires / follow instructions during fMRI assessments and aiTBS treatments. Stated willingness to comply with all study procedures, including availability for the duration of the study, and to communicate with study personnel about adverse events and other clinically important information.
4. Currently diagnosed with either Major Depressive Disorder (MDD) and meets criteria for a current Major Depressive Episode (MDE) according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5).
5. Medical records confirming a history of moderate to severe treatment-resistance as defined by a score of 7-14 on the Maudsley Staging Method (MSM).
6. Endorses clinically significant explicit suicidal cognitions (score ≥ 9 on the M-SSI and score ≥ 6 on the BSS self-report) at screening.
7. MADRS score of >/=20 at screening (visit 1).
8. rTMS/iTBS naive.
9. Access to ongoing psychiatric care before and after completion of the study.
10. Access to clinical rTMS after hospital discharge.
11. In good general health, as evidenced by medical history.
12. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.
13. Agreement to adhere to Lifestyle considerations:

    * Abstain from becoming pregnant from the screening visit (Visit 1) until after the final study visit (Visit 9).
    * Abstain from caffeine- or xanthine-containing products (e.g., coffee, tea, cola drinks, and chocolate) for 3 hours before the start of each dosing session until after the final TMS session.
    * Abstain from alcohol for 24 hours before the start of each dosing session until after collection of the final MRI.
    * Participants who use tobacco products will be instructed that use of cigarettes will not be allowed during the trial.

Exclusion Criteria:

1. Females who are pregnant or planning to become pregnant during the course of the study or any female that is breastfeeding
2. The presence or diagnosis of prominent anxiety disorder, personality disorder, or dysthymia in which in the Investigator's opinion is predominant to MDD
3. Depressed mood/dysphoria as a result of an illness other than MDD (e.g. gender dysphoria)
4. Current severe insomnia (must sleep a minimum of 5 hours each night before stimulation)
5. Current mania or psychosis
6. Bipolar Affective Disorder I and primary psychotic disorders.
7. Autism Spectrum disorder or Intellectual Disability
8. A diagnosis of obsessive-compulsive disorder (OCD)
9. Current moderate or severe substance use disorder or demonstrating signs of acute substance withdrawal.
10. Urine screening test positive for illicit substances.
11. Any history of ECT (greater than 8 sessions) without meeting responder criteria
12. No recent (during the current depressive episode) or concurrent use of a rapid acting antidepressant agent (i.e., ketamine or a course of ECT).
13. History of significant neurologic disease, including dementia, Parkinson's or Huntington's disease, brain tumor, unexpected seizure/epilepsy disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma.
14. Untreated or insufficiently treated endocrine disorder.
15. Contraindications to receiving rTMS (e.g., metal in head, history of seizure, known brain lesion)
16. Contraindications to MRI (ferromagnetic metal in their body).
17. Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.
18. Treatment with another investigational drug or other intervention within the study period.
19. Depth-adjusted SAINT® treatment dose > 65% maximum stimulator output (MSO)
20. Any other condition deemed by the PI to interfere with the study or increase risk to the participant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Change in the neural network underlying Explicit Suicidal Cognition (ESC) as measured by resting state functional connectivity changes in subgenual anterior cingulate (sgACC) and the default mode network (DMN). | At baseline (day 0) and at post-inpatient treatment completion (day 2-7)
  We will assess resting state functional connectivity between sgACC and the DMN and within the DMN using magnetic resonance imaging.

SECONDARY OUTCOMES:
Change in the neural network underlying Implicit Suicidal Cognition (ISC) as measured by resting state functional connectivity changes in dorsolateral prefrontal cortex (DLPFC) and the anterior cingulate cortex (ACC). | At baseline (day 0) and at post-inpatient treatment completion (day 2-7)
  We will use resting state functional connectivity of DLPFC to the ACC using magnetic resonance imaging.

OTHER OUTCOMES:
Change in the neural networks underlying depression, hopelessness and anhedonia as measured by resting state functional connectivity changes of sgACC and medial orbitofrontal cortex (mOFC). | At baseline (day 0) and at post-inpatient treatment completion (day 2-7)
  We will use resting state functional connectivity of sgACC to the mOFC using magnetic resonance imaging to assess connectivity patterns correlated with hopelessness.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Bentzley, MD, Study Director — Magnus Medical
Locations (4):
- United States (4):
  - University of Iowa, Iowa City, Iowa
  - Weill Cornell Medicine, Manhattan, New York
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - University of Texas, Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] Pascual-Leone A, Rubio B, Pallardo F, Catala MD. Rapid-rate transcranial magnetic stimulation of left dorsolateral prefrontal cortex in drug-resistant depression. Lancet. 1996 Jul 27;348(9022):233-7. doi: 10.1016/s0140-6736(96)01219-6. PMID 8684201
- [Background] Abdallah CG, Averill LA, Collins KA, Geha P, Schwartz J, Averill C, DeWilde KE, Wong E, Anticevic A, Tang CY, Iosifescu DV, Charney DS, Murrough JW. Ketamine Treatment and Global Brain Connectivity in Major Depression. Neuropsychopharmacology. 2017 May;42(6):1210-1219. doi: 10.1038/npp.2016.186. Epub 2016 Sep 8. PMID 27604566
- [Background] Liston C, Chen AC, Zebley BD, Drysdale AT, Gordon R, Leuchter B, Voss HU, Casey BJ, Etkin A, Dubin MJ. Default mode network mechanisms of transcranial magnetic stimulation in depression. Biol Psychiatry. 2014 Oct 1;76(7):517-26. doi: 10.1016/j.biopsych.2014.01.023. Epub 2014 Feb 5. PMID 24629537
- [Background] Green KL, Brown GK, Jager-Hyman S, Cha J, Steer RA, Beck AT. The Predictive Validity of the Beck Depression Inventory Suicide Item. J Clin Psychiatry. 2015 Dec;76(12):1683-6. doi: 10.4088/JCP.14m09391. PMID 26717528
- [Background] Ballard ED, Reed JL, Szczepanik J, Evans JW, Yarrington JS, Dickstein DP, Nock MK, Nugent AC, Zarate CA Jr. Functional Imaging of the Implicit Association of the Self With Life and Death. Suicide Life Threat Behav. 2019 Dec;49(6):1600-1608. doi: 10.1111/sltb.12543. Epub 2019 Feb 13. PMID 30761601
- [Background] Tello N, Harika-Germaneau G, Serra W, Jaafari N, Chatard A. Forecasting a Fatal Decision: Direct Replication of the Predictive Validity of the Suicide-Implicit Association Test. Psychol Sci. 2020 Jan;31(1):65-74. doi: 10.1177/0956797619893062. Epub 2019 Dec 11. PMID 31825760
- [Background] Light SN, Bieliauskas LA, Taylor SF. Measuring change in anhedonia using the "Happy Faces" task pre- to post-repetitive transcranial magnetic stimulation (rTMS) treatment to left dorsolateral prefrontal cortex in Major Depressive Disorder (MDD): relation to empathic happiness. Transl Psychiatry. 2019 Sep 3;9(1):217. doi: 10.1038/s41398-019-0549-8. PMID 31481688
- [Background] Baeken C, Duprat R, Wu GR, De Raedt R, van Heeringen K. Subgenual Anterior Cingulate-Medial Orbitofrontal Functional Connectivity in Medication-Resistant Major Depression: A Neurobiological Marker for Accelerated Intermittent Theta Burst Stimulation Treatment? Biol Psychiatry Cogn Neurosci Neuroimaging. 2017 Oct;2(7):556-565. doi: 10.1016/j.bpsc.2017.01.001. Epub 2017 Jan 20. PMID 29560909
- [Background] Downar J, Geraci J, Salomons TV, Dunlop K, Wheeler S, McAndrews MP, Bakker N, Blumberger DM, Daskalakis ZJ, Kennedy SH, Flint AJ, Giacobbe P. Anhedonia and reward-circuit connectivity distinguish nonresponders from responders to dorsomedial prefrontal repetitive transcranial magnetic stimulation in major depression. Biol Psychiatry. 2014 Aug 1;76(3):176-85. doi: 10.1016/j.biopsych.2013.10.026. Epub 2013 Nov 28. PMID 24388670
- [Background] Duprat R, De Raedt R, Wu GR, Baeken C. Intermittent Theta Burst Stimulation Increases Reward Responsiveness in Individuals with Higher Hedonic Capacity. Front Hum Neurosci. 2016 Jun 16;10:294. doi: 10.3389/fnhum.2016.00294. eCollection 2016. PMID 27378888
- [Background] Schmaal L, van Harmelen AL, Chatzi V, Lippard ETC, Toenders YJ, Averill LA, Mazure CM, Blumberg HP. Imaging suicidal thoughts and behaviors: a comprehensive review of 2 decades of neuroimaging studies. Mol Psychiatry. 2020 Feb;25(2):408-427. doi: 10.1038/s41380-019-0587-x. Epub 2019 Dec 2. PMID 31787757
- [Background] Gartner M, Aust S, Bajbouj M, Fan Y, Wingenfeld K, Otte C, Heuser-Collier I, Boker H, Hattenschwiler J, Seifritz E, Grimm S, Scheidegger M. Functional connectivity between prefrontal cortex and subgenual cingulate predicts antidepressant effects of ketamine. Eur Neuropsychopharmacol. 2019 Apr;29(4):501-508. doi: 10.1016/j.euroneuro.2019.02.008. Epub 2019 Feb 26. PMID 30819549